CLINICAL TRIAL: NCT04486898
Title: Effect of Music Therapy in Relieving Burnout Among Nurses
Brief Title: Music Therapy on Burnout Reduction in Nurses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Hsiao-Yean Chiu, Associate Professor, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB 2020-002
Record Dates: First submitted 2020-07-21; First posted 2020-07-27 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Burnout
Keywords: nurses, music therapy,
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Intervention Model Description: This will be a randomized controlled trial with single-blinded, two-arm parallel study. Data will be collected between August to December 2020. A structured questionnaire will be used to collect data on demographics, burnout, depression, stress, and anxiety. We will enroll nurses from the General units of Leroj Atama Memorial Hospital in Majuro, Marshall Islands. The invitation to participate will be communicated by the Chief Nursing Officer and baseline assessment will be given by a trained study interviewer for participant recruitment
Who Masked: Outcomes Assessor
Masking Description: The participants and treatment provider are aware of group assignment due to the nature of biobehavioral intervention. A single-blinded design will be adopted because outcome assessors will be blinded to the group allocation and interventions employed in the two groups. The outcome assessors will not be allowed to disclose participant grouping or to discuss the details of participants. The researcher will not discuss participant-related research data with the outcome assessors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music group (Experimental): Music group will be receiving music intervention 3 times a day for 30 minutes per session for the duration of five (5) weeks period.
  Interventions: Other: Music group
- Usual care (No Intervention): Those who will be in this group will be ask to continue doing their actual activities and not to partake in any kind of music listening or therapy for the 5 week period.

INTERVENTIONS:
Other: Music group — Music group will be given music intervention or listen to music for 30 minutes ,3 times a week for the period of 5 week duration. Music will be selected as per participant's preference
  Arms: Music group

SUMMARY:
This study aims to investigate the effects of music intervention in relieving burnout among nurses. Burnout is a condition of deceased job performance resulting from increased stress in the workplace.This study is to attempt to examine whether music therapy would decrease burnout symptoms and whether there would be a greater decrease of burnout in the music intervention group than the non-music intervention group. In this randomized controlled trial study, we will be using a convenience sample of nurses from Emergency room, medical unit, surgical unit, pediatric, ICU, labor and delivery at the Majuro hospital. Participant will be met for three session each week for a five week period. The participant will be divided into an experimental group (group A) using a music relaxation intervention and control group (group B) with usual care. The study will used the Maslach Burnout Inventory (MBI) with a pretest/post-test design measuring burnout at the beginning before the first session starts and at the end of the last session ends. We hypothesized that clinical nurses who will received music intervention will experience reduction in burnout compared with those in control group will not.

DETAILED DESCRIPTION:
We aim to explore the potential of music therapy to support burnout among nurses and convenience sampling method will be adopted. This will be a randomized single-blinded, two-arm, parallel study, with data to be collected between August to December 2020. Eligible participants will be assigned to either music therapy group or the waiting-list control group. This study will be submitted to Leroj Atama Memorial Hospital at the Ministry of Health and Human Services and the College of the Marshall Islands Research committee for approval.We will enroll nurses from the General units of Leroj Atama Memorial Hospital in Majuro, Marshall Islands. The invitation to participate will be communicated by the Chief Nursing Officer and baseline assessment will be given by a trained study interviewer for participant recruitment. A structured questionnaire will be used to collect data on demographics, burnout, depression, stress, and anxiety. Participants will be recruited from the emergency units and 5 inpatients wards of general hospital of Leroj Atama Memorial Hospital in Majuro, Marshall Islands. We anticipate to enroll 42 nurses into this study. They will be divided into 2 group which are 21 for music group and 21 for control group.Random assignment will be performed by generating sequential numbers using computer software. The random sequential number will then be sealed in thick, opaque, consecutively numbered envelopes before data collections by an independent investigator. Patients will be allocated to either intervention or control group depending on the sequences number revealed by principal investigator. all participants in the music group will receive music intervention over five weeks. Each participant receives music intervention 30 mins per session (2 pm or 4 pm), three days in a week according to their schedule. Music intervention will be conducted at a quiet environment (i.e., nursing lounge) in the hospital. Four types of music protocols based on different rhythm or tones will provide to them, such as classical, slow music, traditional, and Christian song, before the session. Participants will listen to the songs selected and be given mp3 and earpiece for delivering the intervention. During each music session, individual will be advised to close his/her eyes and relaxed and only think of a happy memory. Participant in the waiting-list control group will be asked to maintain their daily routine and they will receive music intervention after the completion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Licensed Registered Nurse
* 3 and more years of work experience
* Complaint of burnout syndrome
* Can speak English
* Consented

Exclusion Criteria:

* diagnosed with advanced cancer

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-11-28 (Actual); Study Completion 2020-11-28 (Actual)

PRIMARY OUTCOMES:
Burnout | at baseline
  Burnout will be measured using Maslach Burnout Inventory questionnaire scale, 22 items subscales of the 3 domain show high consistency with Cronbach's α coefficient values of 0.837, 0.869, and 0.881 and test-retest reliability was high ( p<0.001 ). At baseline, we will collect data regarding burnout level, depression, anxiety, stress and demographic characteristic ( i.e, age, gender, marital status, and having children ect. ) that have been demonstrated to be associated with nurse burnout. The outcome indicators will be collected at 5 weeks after the completion of the intervention. Respondents in the waiting-list control group will complete self-report measures at the same time points as those in the music intervention group.
Burnout | the 5th week after the treatment completion
  Burnout will be measured using Maslach Burnout Inventory questionnaire scale, 22 items subscales of the 3 domain show high consistency with Cronbach's α coefficient values of 0.837, 0.869, and 0.881 and test-retest reliability was high ( p<0.001 ). At baseline, we will collect data regarding burnout level, depression, anxiety, stress and demographic characteristic ( i.e, age, gender, marital status, and having children ect. ) that have been demonstrated to be associated with nurse burnout. The outcome indicators will be collected at 5 weeks after the completion of the intervention. Respondents in the waiting-list control group will complete self-report measures at the same time points as those in the music intervention group.

SECONDARY OUTCOMES:
Depression, anxiety and stress | at baseline
  They will be measured using a self-reported questionnaire, the 21-item Depression Anxiety Stress Score scale (DASS). It assesses the autonomic arousal, skeletal muscle effects, situational anxiety and subjective experience of anxious for anxiety scale, depression scale assesses dysphoria, hopelessness, devaluation of life, self-deprecation, lack of interest/involvement, anhedonia, and inertia, and stress scale assesses difficulty relaxing, nervous arousal, and being easily upset/agitated, irritable and impatient. Subjects are asked to use 4-point scale from 0 'do not apply to me at all' to 3 'apply to me very much' severity/frequency to rate the extent to which they have experienced each state over the past week, DASS score are calculated by summing the scores for the relevant items and 11 score or higher indicates probable presence of greater mood disorder. The subdomain score of 28 and above indicates extremely severe of depression level; the score of 20 and above reflects extremely
Depression, anxiety and stress | the 5th week after the treatment completion
  They will be measured using a self-reported questionnaire, the 21-item Depression Anxiety Stress Score scale (DASS). It assesses the autonomic arousal, skeletal muscle effects, situational anxiety and subjective experience of anxious for anxiety scale, depression scale assesses dysphoria, hopelessness, devaluation of life, self-deprecation, lack of interest/involvement, anhedonia, and inertia, and stress scale assesses difficulty relaxing, nervous arousal, and being easily upset/agitated, irritable and impatient. Subjects are asked to use 4-point scale from 0 'do not apply to me at all' to 3 'apply to me very much' severity/frequency to rate the extent to which they have experienced each state over the past week, DASS score are calculated by summing the scores for the relevant items and 11 score or higher indicates probable presence of greater mood disorder. The subdomain score of 28 and above indicates extremely severe of depression level; the score of 20 and above reflects extremely

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Molina-Praena J, Ramirez-Baena L, Gomez-Urquiza JL, Canadas GR, De la Fuente EI, Canadas-De la Fuente GA. Levels of Burnout and Risk Factors in Medical Area Nurses: A Meta-Analytic Study. Int J Environ Res Public Health. 2018 Dec 10;15(12):2800. doi: 10.3390/ijerph15122800. PMID 30544672